CLINICAL TRIAL: NCT06570720
Title: ASSIST Study: Pilot Cluster Randomized Trial
Brief Title: Alcohol-focused Support of Survivors in Sororities Training (ASSIST) - Pilot
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Washington (Other)
Collaborators: National Institute on Alcohol Abuse and Alcoholism (NIAAA) (NIH)
Responsible Party: Principal Investigator, Anna Jaffe, Associate Professor, Department of Psychiatry and Behavioral Sciences, University of Washington
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: STUDY00018662; K08AA028546 (NIH)
Record Dates: First submitted 2024-08-14; First posted 2024-08-26 (Actual); Last update posted 2025-02-19 (Actual); Status verified 2025-02

CONDITIONS: Alcohol Drinking in College
MeSH Terms: conditions — Alcohol Drinking in College | interventions — Ethanol; Insemination, Artificial, Heterologous

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- ASSIST (Experimental): Participants in this arm will receive online survey assessments as well as the behavioral intervention, ASSIST.
  Interventions: Behavioral: Alcohol-focused Support of Survivors in Sororities Training (ASSIST)
- Assessment-Only (No Intervention): Participants in this arm will only receive online survey assessments.

INTERVENTIONS:
Behavioral: Alcohol-focused Support of Survivors in Sororities Training (ASSIST) — A web-based intervention that includes sorority and individual values, personalized normative feedback (adapted to address sexual assault, support, and acceptability of encouraging peer drinking), psychoeducation on sexual assault and alcohol, and skills training in behaviors to support sexual assault survivors without heavy drinking.
  Arms: ASSIST

SUMMARY:
The goal of this clinical trial is to conduct a preliminary evaluation of the ASSIST (Alcohol-focused Support of Survivors in Sororities Training) intervention in sorority chapters. ASSIST is a newly developed web-based intervention to increase peer support of sexual assault survivors and reduce encouragement of drinking to cope within social networks of sororities. To test whether the intervention is feasible and shows preliminary signs of working, a pilot cluster randomized trial will be conducted. Sorority chapters will be recruited and randomly assigned to an intervention condition or an assessment-only condition. Individuals within each sorority will be recruited and complete a norm documentation survey. One month later, participants will complete a baseline survey, and if assigned to the intervention condition, will then receive the web-based ASSIST intervention, which will include normative feedback on values and drinking, psychoeducation about sexual assault recovery and the role of alcohol, and skills training in behaviors that can be used to support survivors without or while moderating heavy drinking. All participants will complete online follow-up surveys at 1-, 3-, and 6-months post-intervention.

ELIGIBILITY:
Chapter-Level Inclusion Criteria:

* Greek organization of undergraduate women recognized by the Office of Fraternity & Sorority Life with a physical house for chapter members
* At least 80 active members

Individual-Level Inclusion Criteria:

* Aged 18 years or older
* Current student
* Active member in a participating sorority chapter

Exclusion Criteria:

* [None]

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Gender Based: Yes — Participant eligibility is based on sorority membership
Enrollment: 600 (Estimated)
Dates: Start 2024-10-18 (Actual); Primary Completion 2026-05-31 (Estimated); Study Completion 2026-06-30 (Estimated)

PRIMARY OUTCOMES:
Perceived helpfulness | Immediate post-intervention
  Participants will rate the helpfulness of information provided. Range: 1 to 5. Higher scores represent greater helpfulness.
Social Support | Baseline; 1-, 3-, and 6-month follow-up
  On the Multidimensional Scale of Perceived Social Support (MSPSS), participants will rate the support of family, friends, and a significant other. A mean score will be computed. Range: 1 to 7. Higher scores represent more social support.
Alcohol use | Baseline; 1-, 3-, and 6-month follow-up
  On the Daily Drinking Questionnaire (DDQ), participants will report how many standard drinks (0 to 25+) they consumed each day for a typical week in the past month. Total number of drinks per week will be calculated. Range: 0 to 175. Higher scores represent more alcohol use.
Alcohol-related consequences | Baseline; 1-, 3-, and 6-month follow-up
  On the Brief Young Adult Alcohol Consequences Questionnaire (B-YAACQ), participants will indicate whether they have experienced each of 24 negative consequences of alcohol use in the past month. A count of number of consequences experienced will be calculated. Range: 0-24. Higher scores represent more consequences experienced.

CONTACTS AND LOCATIONS:
Overall Officials: Anna Jaffe, Principal Investigator — University of Washington
Locations (1):
- University of Washington, Seattle, Washington, United States

IPD SHARING:
Plan to Share IPD: No